CLINICAL TRIAL: NCT05475106
Title: Pilot Study of Personalized Neoantigen Peptide Vaccines and Leukine for the Treatment of Neoplasms
Brief Title: Pilot Study of Neoantigen Peptides and Leukine for the Treatment of Neoplasms
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Instituto de Medicina Regenerativa (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP-NEO-002
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-01

CONDITIONS: Neoplasms
Keywords: tumor; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients will receive intradermal injection of individualized neoantigen peptides vaccine at a dose of ~500ug per peptide once a week for 4 weeks and once every month after that for 5 months.
  Interventions: Biological: Neoantigen Peptides

INTERVENTIONS:
Biological: Neoantigen Peptides — Patients will receive intradermal injection of individualized neoantigen peptides vaccine at a dose of ~500ug per peptide once a week for 4 weeks, and every month for 5 months after that.

SUMMARY:
The present study is a pilot clinical trial using personalized neoantigen peptide vaccines with the addition of Leukine (Sargramostim), in patients with different types of cancer.

DETAILED DESCRIPTION:
Rationale: Cancer cells express unique peptide antigens recognized by CD8+ cytotoxic T lymphocytes (CTL), which are typically 8-10 amino acids long and are presented in association with Class I MHC molecules. The peptides recognized by helper (CD4+) T-cells are presented in association with Class II MHC molecules and are usually longer (13-18 amino acids in length), although peptide elution studies have indicated no apparent restriction on peptide length. Selected peptides can induce circulating T cell responses in most patients, and that vaccination with a mixture of peptides is immunogenic in up to 100% of patients. The magnitude of T cell responses sometimes is substantial, with 1-5% of circulating CD8 T cells reactive to single antigens. T cell responses to vaccines may be durable for months or years, but are at least as likely to be transient, sometimes declining even while still receiving vaccines. However, T cells induced by vaccination can recognize and lyse cancerous cells expressing the relevant protein and MHC, and peptide vaccines induce promising immunogenicity.

Though MHC-restriction of individual peptides limits their use to a subset of patients, there are mixtures of a dozen peptides restricted by HLA-A1, A2, A3, or A11 can be prepared as a stable mixture and can induce immune responses in 85% of patients with cancer who express one or more of those MHC molecules, without negative effects from competition among the peptides. Other experience supports the ability to induce T cell responses to multiple peptides when vaccinating with peptide mixtures. Since antigenic peptides are easily degraded by proteases in the body, it is difficult for the receptors expressed on the immune cells to identify antigen epitopes, and they do not generate a strong immune response to pathogens. An epitope-based vaccine with a reasonable design is composed of epitope peptide/s, and a delivery system. For multi-epitope vaccines, since the traditional carriers and adjuvants are associated with poor efficacy, vaccine designs with built-in adjuvants have been proposed. Therefore, a built-in adjuvant exhibiting both the functions of a transmission system and a traditional adjuvant, is constructed within the vaccine to improve the immunogenicity of epitope peptides by stimulating the innate immune response required for an adaptive immune response. To achieve this goal, the epitopes are regularly fused with adjuvant proteins or displayed on the surface of some particular biomaterials (e.g., liposomes, gold nanoparticles, and poly(lactic-co-glycolic acid) (PLGA)) and the immunogenicity of the epitopes are significantly increased by this immune complex.

Leukine is the first and only FDA-approved GM-CSF that supports the survival, growth, and activation of neutrophils, monocytes, macrophages, and myeloid-derived dendritic cells. It boosts and stimulate T cells, promoting tissue repair and wound healing, mediating defense against fungal and bacterial pathogens, and producing anti- and pro-inflammatory cytokines, it also improves dendritic cell activity, which is responsible for antigen presentation and immune response regulation. This symbiotic activity potentiates the action of the peptide vaccine.

Study design: This research is a pilot clinical trial using a personalized neoantigen peptide vaccine. Approximately 100 patients with cancer and whose sequencing studies show the presence of neoantigens will receive the personalized multi-peptide vaccine. Peptide vaccines will be given with the addition of Leukine (Sargramostim 250 mcg/m2/dose) by intradermal injection (~0.5 mg of each peptide) in the arm every week for 4 weeks and once every month thereafter for 5 months; the treatment will be discontinued if disease progresses or if there is deterioration of the patient's general condition. All patients will give written informed consent; their data will be coded and fully anonymized. The study was approved by the Ethics Committee of the Regenerative Medicine Institute and conformed to the ethical guidelines of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older, male or female
* Life expectancy of at least 3 months
* Confirmed tumor by imaging studies
* Have adequate organ function, as measured by laboratory values: Lymphocyte ratio >20%; WBC >3.0×10^9/L; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN; if the patient has liver metastases, ALT and AST ≤5 × ULN; Alkaline phosphatase (ALP）≤2.5 × ULN; total serum bilirubin (TBIL) < 1.5 × ULN; Urea nitrogen (BUN）≤1.5 × ULN; Creatinine (Cr）1.5≤ULN; Normal blood coagulation function, urine routine, and electrocardiogram (ECG)
* Available tumor specimen for sequencing and neoantigen determination
* Ability to find 3 or more neoantigen epitopes
* Ability to follow research and follow-up procedures
* Able to understand and willing to sign an IRB approved written informed consent document
* Agree with the use of contraception or partner of child-bearing potential agrees to use adequate contraception which will include two of the following: hormonal or barrier method of birth control, or abstinence prior to study entry, for the duration of study participation, and for 30 days following completion of therapy

Exclusion Criteria:

* History of immunodeficiency disorder or autoimmune condition requiring active immunosuppressive therapy
* Evidence of Liver and kidney dysfunction, severe heart disease, or coagulation dysfunction
* Known diagnosis of an infectious condition including hepatitis, HIV, CMV, and Treponema pallidum
* Participant becomes pregnant and/or is breastfeeding or plans on becoming pregnant during study
* A psychiatric illness that would limit compliance with study requirements as determined by the investigator or the investigator believes that participant is not suitable for inclusion

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in WBC count | Baseline, 2, 6, 12 months
  WBC quantification in blood and comparison at different timepoints
Change from Baseline in RBC count | Baseline, 2, 6, 12 months
  RBC quantification in blood and comparison at different timepoints

SECONDARY OUTCOMES:
Change from Baseline in Calcitonin levels | Baseline, 2, 6, 12 months
  Measured in blood, to assess treatment response at different timepoints
Change from Baseline in CA-125 levels at | Baseline, 2, 6, 12 months
  Measured in blood, to assess treatment response at different timepoints
Change from Baseline in beta-2-microglobulin levels | Baseline, 2, 6, 12 months
  Measured in blood and urine, to assess treatment response at different timepoints
Change from Baseline in sum of diameter of target lesions | Baseline, 2, 6, 12 months
  Measured in the longest diameter in the plane of measurement in CT according to RECIST 1.1 criteria
Change from Baseline in sum of diameter of non-target lesions | Baseline, 2, 6, 12 months
  Measured in the longest diameter in the plane of measurement in CT according to RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Perez, MD, Principal Investigator — Principal Investigator
Locations (1):
- Instituto de Medicina Regenerativa, Tijuana, Estado de Baja California, Mexico